CLINICAL TRIAL: NCT07376343
Title: Comparative Study of CPAP Predictive Equations and In-laboratory Manual Titration in Thai Patients With Obstructive Sleep Apnea
Status: Not yet recruiting | Type: Observational
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Narongkorn Saiphoklang, MD, Associate Professor, Thammasat University
Other Study IDs: TUH-EC-OO-0-031/68
Record Dates: First submitted 2026-01-17; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: OSA - Obstructive Sleep Apnea
Keywords: OSA; obstructive sleep apnea; CPAP; continuous positive airway pressure; equation; Thailand; sleep test; polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obstructive sleep apnea (OSA): Patients aged 18 years or older with OSA
  Interventions: Diagnostic Test: Sleep test; Other: Predictive equations of continuous positive airway pressure (CPAP)

INTERVENTIONS:
Diagnostic Test: Sleep test — Type 1 polysomnography will be performed in the Sleep Center of Thammasat (SCENT).
Other: Predictive equations of continuous positive airway pressure (CPAP) — CPAP predictive equations will be selected based on evidence from reliable studies.

SUMMARY:
The goal of this observational study is to compare predictive equations for continuous positive airway pressure (CPAP) with in-laboratory manual titration in patients with obstructive sleep apnea (OSA).

The main question the study aims to answer is:

Which CPAP predictive equation best predicts the optimal CPAP pressure in OSA patients in Thailand? Participants will undergo an in-laboratory sleep study.

DETAILED DESCRIPTION:
This study is a cross-sectional study involving Thai patients aged 18 years or older with suspected obstructive sleep apnea (OSA). Participants will undergo an in-laboratory sleep study. During the study, sleep technicians will use CPAP predictive equations to estimate the optimal CPAP pressure.

ELIGIBILITY:
Inclusion Criteria:

* Suspected OSA
* Undergoing an in-laboratory sleep study

Exclusion Criteria:

* No indication for in-laboratory manual CPAP titration
* Failure to determine an optimal CPAP pressure during in-laboratory manual CPAP titration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older with suspected OSA
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of CPAP equations in predicting the optimal pressure in OSA patients | At baseline
  Sensitivity and specificity (%) of CPAP equations in predicting the optimal pressure in OSA patients

CONTACTS AND LOCATIONS:
Overall Officials: Narongkorn Saiphoklang, Principal Investigator — Thammasat University Faculty of Medicine
Locations (1):
- Faculty of Medicine, Thammasat University, Pathum Thani, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Yes
IPD and documents will be available for sharing immediately after publication for a period of 2 years.
Supporting Information: Study Protocol, SAP
Time Frame: IPD and documents will be available for sharing immediately after publication for a period of 2 years.

REFERENCES:
- [Result] Lin IF, Chuang ML, Liao YF, Chen NH, Li HY. Predicting effective continuous positive airway pressure in Taiwanese patients with obstructive sleep apnea syndrome. J Formos Med Assoc. 2003 Apr;102(4):215-21. PMID 12833183
- [Result] Chuang ML, Lin IF, Vintch JR, Liao YF. Predicting continuous positive airway pressure from a modified split-night protocol in moderate to severe obstructive sleep apnea-hypopnea syndrome. Intern Med. 2008;47(18):1585-92. doi: 10.2169/internalmedicine.47.1107. Epub 2008 Sep 16. PMID 18797117
- [Result] Luo J, Xiao S, Qiu Z, Song N, Luo Y. Comparison of manual versus automatic continuous positive airway pressure titration and the development of a predictive equation for therapeutic continuous positive airway pressure in Chinese patients with obstructive sleep apnoea. Respirology. 2013 Apr;18(3):528-33. doi: 10.1111/resp.12014. PMID 23145885
- [Result] Wu MF, Hsu JY, Huang WC, Shen GH, Wang JM, Wen CY, Chang KM. Should sleep laboratories have their own predictive formulas for continuous positive airway pressure for patients with obstructive sleep apnea syndrome? J Chin Med Assoc. 2014 Jun;77(6):283-9. doi: 10.1016/j.jcma.2014.02.015. Epub 2014 Apr 14. PMID 24731756
- [Result] Pang F, Deng W, Huang J, Guo Y, Lin M, Zhang X, Liu J. Prediction of Optimal Positive Airway Pressure in Chinese Patients With Obstructive Sleep Apnea. Clin Respir J. 2024 Dec;18(12):e70047. doi: 10.1111/crj.70047. PMID 39716408
- [Result] Choi JH, Kim EJ, Kim KW, Choi J, Kwon SY, Lee HM, Kim TH, Lee SH, Shin C, Lee SH. Optimal continuous positive airway pressure level in korean patients with obstructive sleep apnea syndrome. Clin Exp Otorhinolaryngol. 2010 Dec;3(4):207-11. doi: 10.3342/ceo.2010.3.4.207. Epub 2010 Dec 22. PMID 21217962
- [Result] Lee GH, Kim MJ, Lee EM, Kim CS, Lee SA. Prediction of optimal CPAP pressure and validation of an equation for Asian patients with obstructive sleep apnea. Respir Care. 2013 May;58(5):810-5. doi: 10.4187/respcare.01860. PMID 23051618
- [Result] Sarma L, Putti N, Alias K, Chilana M. Determination of equation for estimating continuous positive airway pressure in patients with obstructive sleep apnea for the Indian population. Lung India. 2020 Sep-Oct;37(5):411-414. doi: 10.4103/lungindia.lungindia_322_19. PMID 32883901
- [Result] Bamagoos AA, Alshaynawi SA, Gari AS, Badawi AM, Alhiniah MH, Alshahrani AA, Rajab RR, Bahaj RK, Alhejaili F, Wali SO. Optimal positive airway pressure requirement and polysomnography indices of obstructive sleep apnea severity in the Saudi population. Ann Thorac Med. 2023 Jan-Mar;18(1):31-38. doi: 10.4103/atm.atm_183_22. Epub 2023 Jan 25. PMID 36968331
- [Result] Ebben MR, Narizhnaya M, Krieger AC. A new predictive model for continuous positive airway pressure in the treatment of obstructive sleep apnea. Sleep Breath. 2017 May;21(2):435-442. doi: 10.1007/s11325-016-1436-7. Epub 2016 Nov 22. PMID 27878543
- [Result] Saiphoklang N, Leelasittikul K, Pugongchai A. Prediction of optimal continuous positive airway pressure in Thai patients with obstructive sleep apnea. Sci Rep. 2021 Jul 6;11(1):13935. doi: 10.1038/s41598-021-93554-5. PMID 34230571